CLINICAL TRIAL: NCT01498042
Title: Ischemic Stroke Treated With iv Thrombolysis Within 4.5 Hours: Predictors of Outcome in a Cohort With a Large Proportion of Patients Above 80 Years
Brief Title: Predictors of Outcome in t-PA Treated Stroke.
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 813387
Record Dates: First submitted 2011-07-06; First posted 2011-12-23 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2011-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stroke, thrombolysis, over 80, outcome: To study the outcome of stroke patients over 80 years treated with thrombolysis.

SUMMARY:
Stroke is among the most disabilitating diseases worldwide in terms of numbers affected and its consequences. A relatively new and well documented treatment of acute ischemic stroke today is tPA (tissue plasminogen activator; will be called thrombolysis from now on) Unfortunately only a minority of patients is given this treatment.

The large randomised controlled trials that investigated the safety and efficacy of thrombolytic therapy in treatment of acute stroke did not include patients over 80 years. In an aging population in the western world it will be of importance to investigate whether this treatment is safe and effective in this group.

Both Sorlandet hospital Kristiansand Norway and Bergen hospital have administered thrombolysis to selected patients over 80 years the last years. In addition there has been a registration of patients in stroke registers at both locations. This lays a foundation for further investigation. In association with Bergen the investigators have included 77 patients over 80 years treated with thrombolysis. In addition the investigators have 85 patients treated with tpa below 80 years. In our cohort the investigators are going to compare outcome in the 2 groups. In addition the investigators are going to perform a regression analysis of selected variables to see if there is an association of those variables with predefined outcome measures. Our outcome measures is as follows: mRS=6 (death)and mRS 0-1(good outcome) on 3 months control. The third outcome measure will be developement of sICH secondary to tPA treatment. As definition of sICH we have chosen the same definition as Ecass.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke treated with thrombolysis over 80 years between 01.01.2007-28.02.2010 from predefined centers.
* Patients with acute ischemic stroke treated with thrombolysis at Sorlandet hospital Kristiansand below 80 years in the same defined period.

Two patients were excluded due to missing data at three months control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sorlandet hospital is a secondary hospital. The patients will be drawn from thrombolysis treated patients in its catchement area. A registry of these patients has been ongoing since before the inclusiondate. All thrombolysed patients at Sorlandet will be included in the predefined inclusionperiode. In addition we have enrolled 39 patients treated with thrombolysis from Haukeland hospital; Bergen. These 77 patients over 80 years will be compared to 85 patients below 80 years treated at SSK in the same defined periode.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Intravenous thrombolysis for acute ischemic stroke with 4.5 hours time-window and no upper age limit | 2007-2010 (3 yrs)
  Functional outcome and complications 3 months after thrombolysis in patients over 80 and under 80 years.

CONTACTS AND LOCATIONS:
Overall Officials: Aase Mygland, MD, PhD, Study Chair — Sørlandet sykehus HF
Locations (1):
- Sørlandet sykehus HF, Kristiansand, Norway